CLINICAL TRIAL: NCT06768502
Title: Effectiveness of Community-based Approach in Reducing the Intimate Partner Violence (IPV) Exposure and Outcome: a Randomized Control Trial of IPV Victimization and Perpetration in Rwanda
Brief Title: Effectiveness of Community-based Approach in Reducing the Intimate Partner Violence (IPV) Exposure and Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rwanda (Other)
Responsible Party: Principal Investigator, Izabayo Josias, Lecturer, University of Rwanda
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMH
Record Dates: First submitted 2024-08-18; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Intimate Partner Violence (IPV); Anxiety; Depression; Post-traumatic Stress Disorder (PTSD)
Keywords: IPV; community support; emotions management; anxiety; depression; PTSD; Rwanda
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: * Arm 1 (Intervention Group): Describe the intervention that this group will receive intervention
  * Arm 2 (Control Group): Describe what the control group will receive no intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): This arm includes couples selected from a list provided by authorities at the sector level, identifying households with a history of family violence. These couples will receive the Community-Based Approach (CBA) intervention and will be assigned to the treatment group.
  Interventions: Other: Community Based Approach (CBA)
- control group (No Intervention): This arm includes couples selected from a list provided by authorities at the sector level, identifying households with a history of family violence. These couples will not receive the Community-Based Approach (CBA) intervention and will be assigned to the control group.

INTERVENTIONS:
Other: Community Based Approach (CBA) — The community-based approach on IPV and sexual violence is conceived as a dynamic process where community members willing to recover from life wounds induced by IPV and sexual violence agree to share their lived experiences in order to work on them accordingly and to support each other in this healing journey.
  Arms: treatment group

SUMMARY:
Abstract

Background:

There is a little known about the effectiveness of Community-Based Approach (CBA) on reduction of intimate partner violence (IPV) exposure, anxiety, depression and PTSD symptoms as outcomes in collectivist and post-genocide societies like Rwanda. This study, therefore, aimed at assessing the effectiveness of Community-Based Approach (CBA) for IPV victimization and perpetration as well as it's associated mental health outcomes in Rwanda.

Methods:

This is a Randomized Controlled Trial (RCT) study which will be conducted using a sample of 31 couples (MA =36.9, SD=9.9), with 16 couples assigned in treatment group and 15 assigned in control group. Data has to be collected using the Hurt, Insult, Threaten and Screaming (HITS-7) to assess IPV exposure; the Hopkins Symptom Checklist for anxiety and depression (HSCL-25); and the PTSD checklist for DSM-5 (PCL-5). Data will be analyzed using Pearson correlation and mixed ANOVAs to evaluate the effect of CBA over IPV occurrence and mental health outcomes.

Key words:

IPV, community support, emotions management, anxiety, depression, PTSD, Rwanda

DETAILED DESCRIPTION:
Introduction Globally, intimate partner violence (IPV) against woman is considered as an important social and public health issue. IPV refers to physical, sexual or emotional harm by a current or former intimate partner. It has been estimated that almost 30% of all women in the world have experienced IPV. South- East Asia, the Mediterranean region and Africa were found to have the highest lifetime prevalence of physical and/or sexual IPV. According to the analysis of data from 77 studies conducted by World Health Organization (WHO), 33% of women have ever experienced physical or sexual violence in Africa region, which was similar to South-East Asia and Mediterranean region (31%). Within the region, the national surveys demonstrated that the prevalence of lifetime physical and/or sexual violence among women from age 15 to 49 years ranges from 47% in Democratic Republic of Congo (DRC) to 16 % in Cameroon . Similarly, the national survey in Rwanda also found that 38% of Rwandan women experience physical and /or sexual violence in their life time which keeps placing Rwanda among the countries with the highest prevalence of intimate partner violence in the world. Recently data from the 2019/2020 Rwanda Demographic and Health Survey(RDHS) has showed that the percentage of women who report IPV experience increased from 40.1% in 2015 to 46% in 2020 but declined from 21% to 17% for men in the same period Exposure to IPV, like any other experiences of violence (gender-based violence, sexual violence), is reported to have deleterious and long-lasting negative effects on the victims. Research findings and clinic records have shown that women who are victims of IPV are likely to report a wide range of negative health consequences (physical and mental) such as depression, anxiety, post-traumatic stress disorder (PTSD), suicide ideations and attempts, alcohol and drug use disorders, physical injuries, and even death.The negative effect of the IPV exposure is reported to affect offspring, meaning that children from families where there is violence may also suffer from a range of behavioral and emotional problems. On the other hand, there is well documented associations between psychopathology and IPV victimization and perpetration. Such comorbidity implies that the association between IPV and mental disorders is bi-directional, meaning that IPV may cause mental sufferance and vice-versa; as such mentally ill individuals are likely to experience or inflict frequent IPV than non-mentally affected individuals.

The genocide committed against Tutsi in Rwanda has left the surviving victims with deep wounds and scars, both physical and mental, which are seen particularly during commemoration events . As from the growing research interests assessing the long-lasting effects of the genocide on both the general population and survivors, results yield quite high prevalence of mental disorders in both samples, with highest scores in the sub-sample of survivors. Equally, scholars estimate the post-traumatic burden to affect not only the direct victims of the genocide but possibly their offspring as well through different mechanisms of transmission. In the same vein, chronic mental disorders, particularly PTSD and depression, are considered to be predictors of the worsening of family harmony and sometimes leading to disputes and related IPV related psychopathologies. In an effort to address IPV and its associated mental health problems being a public health concern in post-genocide Rwanda, some NGOs have developed and implemented programs aimed at empowering women and changing community norms that support violence and male dominance in sub-Saharan Africa. These programs are reported to have had a positive effect on IPV victimization and perpetration with additional intervention benefits like improvement in depression symptoms, conflict management, communication, trust, self-efficacy, household earnings, food security and actions to prevent IPV. Such programs have focused on raising awareness on domestic violence and intimate partner violence, with a working hypothesis that the increase of knowledge on the IPV phenomenon will reduce its perpetration and victimization. Moreover, these studies were limited in their design as few interventions worked on past-mental burden which is likely to negatively affect couples' communication and intimacy. Equally, little attention was directed to the anxiety and PTSD disorders which were estimated to be ubiquitous to IPV exposure and perpetration.

However, amongst the local organizations intervening in the area of domestic violence in Rwanda, the Life Wounds Healing Association (LIWOHA) has almost twenty years' experience of intensive work in communities managing IPV from a Community Based Approach (CBA) by integrating psychoeducation, psychosocial support and emotions management models. The working paradigm of the organisation is that violent behaviours in couples are induced by life wounds rooted in the past. Therefore, unless perpetrators and victims discover the real cause of their violent behaviours and work on them, it assumed that awareness raising and law enforcement themselves will not discourage IPV perpetrators.

In a longitudinal study design examining the impact of the LIWOHA group-based intervention, revealed that the approach was effective in bringing together members of opposing groups (survivors and perpetrators of the genocide) by facilitating mutual healing and restored trust; establishing new social identities, and regained a strong sense of belonging. While this approach is being utilized in managing IPV cases, none of the existing studies have assessed it's effectiveness in lowering IPV perpetration and victimization occurrence as well as it's improvement in outcomes like anxiety, depression, and PTSD symptoms.

Therefore, the aim of this study is to evaluate the effectiveness of the community-based approach in managing IPV, anxiety, depression and PTSD among individuals reporting IPV.

Methods Participants

Participants are to be recruited from Ntungamo and Kankuba cells in Mageragere Sector, City of Kigali. From a list submitted by the Sector Executive Secretary of 113 couples considered by the local authorities as conflicting couples, 58 couples from both cells were eligible for this study. Eligibility criteria included the consent, experience of IPV and availing time to attend all the workshop sessions. Couples accepting to participate in the research were randomly distributed in treatment and control groups. Given number of eligible participants (58 couples), and the need to reduce the number of couples to 15 for both groups, the "first come, first served" principle was used. As such, 32 couples, 17 from Nkankuba Cell (Treatment group) and 15 couples from Ntungamo Cell (control group) granted their consent to participate in the research either as experimental or control.

Procedure

Experimental group will receive the LIWOHA workshops package delivered by a clinical psychologist working with the organization. It will be important that the sessions are facilitated by the same trained staff from the organization to ensure accuracy and fidelity. The workshops structure will take13 days, with time interval of 3 to 4 weeks between sessions. The interval time will mean for participants to practice what they will learn from the preceding session. Structured interviews were conducted in each workshop for the experimental group. On the side of the control group, which did not receive the LIWOHA package, participants were also assessed at the same time as the experimental group. The control group will only be followed and supported by the cells personnel by educating participants on the existing laws and policies for mitigating and punishing all IPV behaviours.

Treatment manualisation

The community-based approach on IPV and sexual violence is conceived as a dynamic process where community members willing to recover from life wounds induced by IPV and sexual violence agree to share their lived experiences in order to work on them accordingly and to support each other in this healing journey. The main steps or sessions of a community healing program can be summarized as follow:

* Awareness and sensitization session (3 days) dedicated to education participants (victims and perpetrators of domestic, gender and sexual violence) on the destructive nature of life wounds rooted in their past as root causes of violent behaviors. The objective of the workshop is to awaken the beneficiaries on the destructive potential of these types of violence as far as family harmony and the social fabric is concerned.
* "Life wounds mourning session" (3 days) dedicated to couples living in permanent conflicts on how to deal accordingly with their important past losses that prevent them from establishing pacified relationships in their families and care for their children (who consequently flee their home, live carelessly, and fall in vulnerability). The objective of this session is to start the healing "journey" that normally results in the re-establishment of harmonious relationships and adoption of positive parenting styles that prevent children from fleeing their home again.
* Sessions dedicated to the "management of negative psychological feelings" (3 days) associated with life wounds. These sessions follow those dedicated to positive mourning and aim at helping beneficiaries to deal accordingly with negative emotions and sentiments induced by life wounds rooted in the past and actual violent behaviors in families.
* Sessions dedicated to "forgiveness and reconciliation with their own past" (2 days) and with others. Workshops related to this step help beneficiaries to reconnect with others. During these sessions, perpetrators of domestic and gender violence ask for forgiveness and make a commitment to no longer abuse their victims and submit themselves to community monitoring.
* The last sessions are dedicated to the "development of a new project for a new life" (2 days). In this last step, healed people define a new lifestyle without violence and commit to resume assuming family responsibilities he/she had abandoned in the past.

Tools

The HITS (Hurt, Insult, Threaten, and Scream) is a 7 items Likert scale which is used to evaluate intimate partner violence. All items were scored as: 0=never, 1=rarely, 2=sometimes, 3=fairly often, and 4=frequently. The total scores ranged from Score 0 to 24.

The Hopkins Symptom Check List-25 is a 25 items instrument which is used to measure common psychiatric symptoms of depression and anxiety in both clinical and non-clinical samples.The first 10 items assess anxiety symptoms and the remaining 15 items assess depression.

The PTSD Checklist (PCL-5) is a 20 items self-reported instrument that was used to evaluate the symptoms of PTSD. All items were scored on the Likert scale: 0=Not at all, 1=A little bit, 2=moderately, 3=Quite a bit and 4=extremely. The total score ranged from 0 to 20.

Ethical consideration

The study was submitted and approved by the University of Rwanda College of Medicine and Health Sciences' Institutional Review Board (IRB); approval letter No 033/CMHS-IRB/2020 of 18th February 2020. Ethical principles were fully complied for and included free informed consent and privacy principles.

Data analysis

Data will be analysed descriptively to describe the characteristics of participants.The effectiveness of community-based approach to victims/perpetrators of Intimate partner violence and mental health disorders will be evaluated using a mixed ANOVAs with a within-subjects' factors and a between-subjects factor. All analysis has to be performed using Statistical Package for Social sciences (SPSS) version 25.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Attended all session

Exclusion Criteria:

* Lost the follow up
* Declined the participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Reduced intimate Partner Violence scores in treatment group as compared to control groups | through study completion, an average of 10 months
  Analysis of effectiveness community based approach in reducing the IPV scores. IPV scores were assessed using The Hurt, Insult, Threaten, and Scream scale which has 7 items with a likert scaled response. All items were scored as: 0=never, 1=rarely, 2=sometimes, 3=fairly often, and 4=frequently. The total scores ranged from Score 0 to 24, where higher scores mean worse outcome.
Reduced Anxiety scores in treatment group as compared to control groups | through study completion, an average of 10 months
  Analysis of effectiveness community based approach in reducing the anxiety scores. The Hopkins Symptom Check List-25 scale was used to evaluate depression scores. Its first 10 items assess anxiety symptoms. The scale for each item includes four categories of response ("Not at all," "A little," "Quite a bit," "Extremely," rated 1 to 4, respectively). The total scores range from 1 to 40, where higher scores mean worse outcome.
Reduced depression scores in treatment group as compared to control groups | through study completion, an average of 10 months
  Analysis of effectiveness community based approach in reducing the depression scores. Its last 15 items assess depression. The scale for each item includes four categories of response ("Not at all," "A little," "Quite a bit," "Extremely," rated 1 to 4, respectively).The total scores range from 1 to 60,where higher scores mean worse outcome.
Reduced post-traumatic stress disorder scores in treatment as compared to control groups | through study completion, an average of 10 months
  Analysis of effectiveness community based approach in reducing post-traumatic stress disorder scores.The PTSD Checklist for DSM-5 (PCL-5) is a 20 items self-reported instrument that was used to evaluate the 20 DSM-5 symptoms of post-traumatic stress disorder (Weathers et al., 2013). All items were scored on the Likert scale: 0=Not at all, 1=A little bit, 2=moderately, 3=Quite a bit and 4=extremely. The total score ranged from 0 to 80, where higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Sezibera, Professor, Principal Investigator — University of Rwanda
Locations (1):
- Centre for Mental Health, Kigali, Western, Rwanda

REFERENCES:
- [Background] Ahmadabadi Z, Najman JM, Williams GM, Clavarino AM, d'Abbs P, Tran N. Intimate partner violence and subsequent depression and anxiety disorders. Soc Psychiatry Psychiatr Epidemiol. 2020 May;55(5):611-620. doi: 10.1007/s00127-019-01828-1. Epub 2020 Jan 7. PMID 31912167
- [Background] Bahati C, Izabayo J, Munezero P, Niyonsenga J, Mutesa L. Trends and correlates of intimate partner violence (IPV) victimization in Rwanda: results from the 2015 and 2020 Rwanda Demographic Health Survey (RDHS 2015 and 2020). BMC Womens Health. 2022 Sep 6;22(1):368. doi: 10.1186/s12905-022-01951-3. PMID 36068627
- [Background] Bahati C, Rukundo G, Nyirahabimana N, Izabayo J, Niyonsenga J, Sezibera V. The prevalence of mental disorders among intimate partner violence exposed and non-exposed Rwandans: Findings from a national cross-sectional survey. Psychiatry Res. 2022 Apr;310:114465. doi: 10.1016/j.psychres.2022.114465. Epub 2022 Feb 19. PMID 35219265
- [Background] Bland JM, Altman DG. Cronbach's alpha. BMJ. 1997 Feb 22;314(7080):572. doi: 10.1136/bmj.314.7080.572. No abstract available. PMID 9055718
- [Background] Bris, T. Le. (2017). The Hopkins symptoms checklist in 25 items : translations in Castilian, Galician, Catalan, French, Greek, Italian, Polish, Bulgarian and Croatian synthesis. Life. Life Science, q-bio, dumas-01537933.
- [Background] Bulte, E. (2020). Empowerment and intimate partner violence : Domestic abuse when household income is uncertain. July, 1-15. https://doi.org/10.1111/rode.12715
- [Background] Celestin, M., Vincent, S., & C, C. (2022). Determinants of Intergenerational Trauma Transmission: A Case of the Survivors of the 1994 Genocide Against Tutsi in Rwanda. Child Behavioral Health in Sub-Saharan Africa. https://doi.org/10.1007/978-3-030-83707-5_11
- [Background] Chatterji, S., & Heise, L. (2021). Examining the bi-directional relationship between intimate partner violence and depression: Findings from a longitudinal study among women and men in rural Rwanda. SSM - Mental Health, 1, 10. https://doi.org/10.1016/j.ssmmh.2021.100038
- [Background] Chilanga E, Collin-Vezina D, Khan MN, Riley L. Prevalence and determinants of intimate partner violence against mothers of children under-five years in Central Malawi. BMC Public Health. 2020 Dec 2;20(1):1848. doi: 10.1186/s12889-020-09910-z. PMID 33267864
- [Background] Clear, T. R. (2007). Imprisoning Communities: How Mass Incarceration Makes Disadvantaged Neighborhoods Worse. https://doi.org/10.1093/acprof:oso/9780195305791.001.0001
- [Background] Davoren, M., Kallis, C., González, R. A., Freestone, M., & Coid, J. W. (2017). Anxiety disorders and intimate partner violence: can the association be explained by coexisting conditions or borderline personality traits? The Journal of Forensic Psychiatry & Psychology. https://doi.org/10.1080/14789949.2016.1172659
- [Background] DeJonghe ES, Bogat GA, Levendosky AA, von Eye A. Women survivors of intimate partner violence and post-traumatic stress disorder: prediction and prevention. J Postgrad Med. 2008 Oct-Dec;54(4):294-300. doi: 10.4103/0022-3859.41435. PMID 18953149
- [Background] Dunkle K, Stern E, Chatterji S, Heise L. Effective prevention of intimate partner violence through couples training: a randomised controlled trial of Indashyikirwa in Rwanda. BMJ Glob Health. 2020 Dec;5(12):e002439. doi: 10.1136/bmjgh-2020-002439. PMID 33355268
- [Background] Dunkle, K., Stern, E., Chatterji, S., Heise, L., Mclean, L., & Chatterji, S. (2019). Indashyikirwa programme to reduce intimate partner violence in Rwanda: Report of findings from a cluster randomized control trial. August, 1-56. https://www.whatworks.co.za/documents/publications/352-indash-evidence-brief-aug-2019/file
- [Background] Esie P, Osypuk TL, Schuler SR, Bates LM. Intimate partner violence and depression in rural Bangladesh: Accounting for violence severity in a high prevalence setting. SSM Popul Health. 2019 Jan 28;7:100368. doi: 10.1016/j.ssmph.2019.100368. eCollection 2019 Apr. PMID 30766911
- [Background] Jabbi A, Ndow B, Senghore T, Sanyang E, Kargbo JC, Bass P. Prevalence and factors associated with intimate partner violence against women in The Gambia: a population-based analysis. Women Health. 2020 Sep;60(8):912-928. doi: 10.1080/03630242.2020.1767264. Epub 2020 May 18. PMID 32419660
- [Background] Kabakambira JD, Uwera G, Hategeka M, Kayitesi ML, Malu CKK, Hategeka C. Burden of post-traumatic stress disorder acute exacerbations during the commemorations of the genocide against Tutsis in Rwanda: a cross-sectional study. Pan Afr Med J. 2018 Jul 17;30:216. doi: 10.11604/pamj.2018.30.216.15663. eCollection 2018. PMID 30574235
- [Background] Kapiga S, Harvey S, Muhammad AK, Stockl H, Mshana G, Hashim R, Hansen C, Lees S, Watts C. Prevalence of intimate partner violence and abuse and associated factors among women enrolled into a cluster randomised trial in northwestern Tanzania. BMC Public Health. 2017 Feb 14;17(1):190. doi: 10.1186/s12889-017-4119-9. PMID 28193198
- [Background] King, R. U. (2019). The true healing is healing together: Healing and rebuilding social relations in postgenocide Rwanda. Peace and Conflict. Journal of Peace Psychology, 25(1), 49-60. https://doi.org/10.1037/pac0000357
- [Background] Lovestad S, Love J, Vaez M, Krantz G. Prevalence of intimate partner violence and its association with symptoms of depression; a cross-sectional study based on a female population sample in Sweden. BMC Public Health. 2017 Apr 20;17(1):335. doi: 10.1186/s12889-017-4222-y. PMID 28424072
- [Background] Musanabaganwa C, Jansen S, Fatumo S, Rutembesa E, Mutabaruka J, Gishoma D, Uwineza A, Kayiteshonga Y, Alachkar A, Wildman D, Uddin M, Mutesa L. Burden of post-traumatic stress disorder in postgenocide Rwandan population following exposure to 1994 genocide against the Tutsi: A meta-analysis. J Affect Disord. 2020 Oct 1;275:7-13. doi: 10.1016/j.jad.2020.06.017. Epub 2020 Jun 23. PMID 32658827
- [Background] Mutuyimana, C., Sezibera, V., & Cassady, C. (2022). Determinants of Intergenerational Trauma Transmission: A Case of the Survivors of the 1994 Genocide Against Tutsi in Rwanda. In F. M. Ssewamala, O. Sensoy Bahar, & M. M. McKay, Child Behavioral Health in Sub-Saharan Africa Towards Evidence Generation and Policy Development (Vols. 213-233). Springer Nature Switzerland AG, Switzerland.
- [Background] Rhodes KV, Houry D, Cerulli C, Straus H, Kaslow NJ, McNutt LA. Intimate partner violence and comorbid mental health conditions among urban male patients. Ann Fam Med. 2009 Jan-Feb;7(1):47-55. doi: 10.1370/afm.936. PMID 19139449
- [Background] Richie, B. E. (2014). Who Benefits and Who Loses in the Criminalization of IPV : Considering the Logic of Punishment and Impact of Legal Intervention as a Tertiary Prevention Strategy. 1-19.
- [Background] Rieder H, Elbert T. Rwanda - lasting imprints of a genocide: trauma, mental health and psychosocial conditions in survivors, former prisoners and their children. Confl Health. 2013 Mar 26;7(1):6. doi: 10.1186/1752-1505-7-6. PMID 23531331
- [Background] Thomson DR, Bah AB, Rubanzana WG, Mutesa L. Correlates of intimate partner violence against women during a time of rapid social transition in Rwanda: analysis of the 2005 and 2010 demographic and health surveys. BMC Womens Health. 2015 Oct 28;15:96. doi: 10.1186/s12905-015-0257-3. PMID 26511348
- [Background] Umubyeyi A, Mogren I, Ntaganira J, Krantz G. Intimate partner violence and its contribution to mental disorders in men and women in the post genocide Rwanda: findings from a population based study. BMC Psychiatry. 2014 Nov 18;14:315. doi: 10.1186/s12888-014-0315-7. PMID 25406929
- [Background] Vindbjerg E, Carlsson J, Mortensen EL, Makransky G, Nielsen T. A Rasch-based validity study of the Harvard Trauma Questionnaire. J Affect Disord. 2020 Dec 1;277:697-705. doi: 10.1016/j.jad.2020.08.071. Epub 2020 Sep 1. PMID 32911220
- [Background] Weathers, F. W., Litz, B. T., Keane, T. M., Palmieri, P. A., Marx, B. P., & & Schnurr, P. P. (2013). The PTSD Checklist for DSM-5 (PCL-5).Scale available from the National Center for PTSD at. www.ptsd.va.gov.
- [Background] Sardinha L, Maheu-Giroux M, Stockl H, Meyer SR, Garcia-Moreno C. Global, regional, and national prevalence estimates of physical or sexual, or both, intimate partner violence against women in 2018. Lancet. 2022 Feb 26;399(10327):803-813. doi: 10.1016/S0140-6736(21)02664-7. Epub 2022 Feb 16. PMID 35182472